CLINICAL TRIAL: NCT06737367
Title: Integrating Machine Learning for Prognostic Prediction in Stage I NSCLC: a Multicenter Analysis
Brief Title: Integrating Machine Learning for Prognostic Prediction in Stage I NSCLC by CT Images and Pathological Factors
Acronym: Stage I NSCLC
Status: Completed | Type: Observational
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Guangming Lu, Professor, Jinling Hospital, China
Other Study IDs: 2023DZKY-089-01
Record Dates: First submitted 2024-12-11; First posted 2024-12-17 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Lung Cancer - Non Small Cell
Keywords: NSCLC, ML, DFS
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- training set
  Interventions: Other: CT radiomic analysis
- external test set
  Interventions: Other: CT radiomic analysis

INTERVENTIONS:
Other: CT radiomic analysis — Radiomic features of tumor and peritumor tissue

SUMMARY:
The investigators retrospectively collected the participants with stage I non-small cell lung cancer (NSCLC) patients resected between January 2010 to December 2020 for training and internal validation. The Clinical data, preoperative clinical information, laboratory results and CT images were collected. The investigators also collected the disease-free survival time. On the Deepwise multi-modal research platform, the images were semi-automatically segmented and expanded outward by 3mm to obtain the peritumor tissue. PyRadiomics was used to extract the radiomic features. LASSOcox and rsf were used to select the features. we developed a machine learning-based integrative prognostic model that utilizes radiomic and pathological variables as input using LOOCV framework. And it was further tested on the internal and external cohorts. Discrimination was assessed by using the C-index and area under the receiver operating characteristic curve (AUC), IBS, DCA.

ELIGIBILITY:
Inclusion Criteria:

patients with stage I NSCLC (ninth AJCC edition) who underwent curative R0 resections between January 2010 and December 2020 -

Exclusion Criteria:

1. absence of enhanced CT
2. history of lung cancer or synchronous lung cancers
3. follow-up records ≤3 Months
4. carcinoma in situ (CIS) or minimally invasive NSCLC
5. death within 30 days of surgery
6. no pathological slides or reports

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Jinling Hospital, China
Sampling Method: Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2024-11-11 (Actual)

PRIMARY OUTCOMES:
DFS（Disease-free survival） | Record from the date of surgery to the date of recurrence or death from any cause, whichever comes first, and assess up to a maximum of 5 years.
  DFS was defined as the duration from the date of primary surgery to the first occurrence of recurrence or death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Jinling Hospital, China, Nanjing, China

IPD SHARING:
Plan to Share IPD: No